CLINICAL TRIAL: NCT07030335
Title: The Effect Of A Mobıle Educatıon Program and Telephone Follow-Up On Knowledge Level, Symptom Management And Qualıty Of Lıfe In Patıents Wıth Atrıal Fıbrıllatıon
Brief Title: Evaluation of Mobile Education Program in Patients With Atrial Fibrillation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Suna Eroğlu Aygül, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AU-İHH-SE-01
Record Dates: First submitted 2025-05-27; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Nursing; Mobile application; Symptom management; Quality of life; Level of knowledge
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Mobile-Atrial Fibrillation Training Program
- Control Group (Placebo Comparator)
  Interventions: Other: Routine Outpatient Clinic Care

INTERVENTIONS:
Other: Mobile-Atrial Fibrillation Training Program — Patient Information Form, Atrial Fibrillation Information Scale, Atrial Fibrillation Severity Scale and Atrial Fibrillation Impact on Quality of Life Questionnaire will be administered face-to-face by the researcher using Mobile Atrial Fibrillation Education Program (M-AFEP). The application link, individual e-mail and user passwords will be sent to the mobile phones of the participants and the application will be added to the main screens by entering the relevant address from their phones. Participants will be asked to use M-AFEP for twelve weeks / at least ten minutes a week and the frequency and duration of use will be recorded on the mobile application. Participants in the intervention group will be followed up by phone once a week in the first, fourth and eighth weeks and a reminder message (sms) will be sent for the use of M-AFEP. At the end of the twelfth week, the scales will be filled in again through the application.
  Arms: Intervention Group
Other: Routine Outpatient Clinic Care — * Participants in the control group will be given M-AFEP application usage training by the researchers.
  * The application link, individual e-mail and user passwords will be sent to the mobile phones of the participants in the control group.
  * Participants in the control group will enter the relevant address of the mobile application from their phones and the application will be added to their home screens.
  * In the M-AFEP application of the participants in the control group, there will be a short general information section containing information specific to AF, different from the intervention group content.
  Participants in the control group will continue only routine outpatient follow-up throughout the process and no intervention will be applied.
  Arms: Control Group

SUMMARY:
This study was conducted to determine the effect of a mobile education program and telephone follow-up on the knowledge level, symptom management and quality of life of patients with atrial fibrillation.

The study aims to answer the following questions.

1. Does the mobile education program and telephone follow-up have an effect on increasing the level of knowledge in patients with AF in the intervention group compared to the control group?
2. Does the mobile education program and telephone follow-up have an effect on reducing symptom severity in patients with AF in the intervention group compared to the control group?
3. Does the mobile education program and telephone follow-up have an effect on improving the quality of life in patients with AF in the intervention group compared to the control group?

DETAILED DESCRIPTION:
The research was planned in two phases: development of the mobile training program and evaluation of its effectiveness. TIn the first phase of the study, M-AFEP (Mobile-Atrial Fibrillation Education Program) application will be developed, and in the second phase of the study, the effectiveness of M-AFEP will be evaluated with a randomized controlled experimental research design with active control group.

The sample of the study will consist of patients diagnosed with AF aged 18 years and older who are followed up for routine controls at the Cardiology Outpatient Clinic of Akdeniz University Hospital and who meet the inclusion criteria.The sample of the study will consist of a total of 70 patients with AF 35 intervention and 35 control groups.

In order to evaluate the comprehensibility of the data collection tools and M-AFEP, it is planned to conduct a four-week pre-application with 4 participants, 10% of the intervention group, before the study. Personal Information Form, Jessa Atrial Fibrillation Knowledge Questionnaire (JAKQ), The University of Toronto Atrial Fibrillation Severity Scale (AFSS), Effect of Atrial Fibrillation on Quality of Life Scale (AFEQT) and System Usability Scale (SUS) will be used for data collection. Participants in the intervention group, whose consent was obtained, will initially be trained on the use of M-AFEP and the M-AFEP application version will be installed on their phones. Then, the researcher will conduct follow-up by telephone in the first, fourth and eighth weeks. Similarly, a reminder message (sms) about the use of M-AFEP will be sent once a week in the first, fourth and eighth weeks.

Participants will use M-AFEP for twelve weeks. At the end of the twelfth week, patients in the intervention and control groups will complete the post-tests (Jessa Atrial Fibrillation Knowledge Questionnaire (JAKQ), The University of Toronto Atrial Fibrillation Severity Scale (AFSS), Effect of Atrial Fibrillation on Quality of Life Scale (AFEQT)) using the mobile application. Participants will evaluate the mobile application with the System Usability Scale. These data will constitute the post-test measurements of the study. After the post-test, the M-AFEP application will be shared with the participants in the control group for their benefit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Being literate.
* Atrial Fibrillation diagnosis.
* No cognitive and communication disabilities.
* Not having a diagnosed psychiatric illness.
* Ability to use technological devices.
* Having and using a smart phone with Android operating system and internet access.
* Acceptance to participate in the study.

Exclusion Criteria:

* Diagnosis of rheumatic valve disease, moderate/severe mitral stenosis and previous valve surgery.
* Functional class III or IV according to the New York Heart Association (NYHA) classification.
* Patients with existing or planned pacemaker, ICD (Implantable Cardioverter Defibrillator) and patients with existing or planned Radiofrequency Ablation treatment will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The Jessa Atrial Fibrillation Knowledge Questionnaire | The measurement will be done at the beginning of the study (day 0) and at the end of the 12th week.
  -The Jessa Atrial Fibrillation Knowledge Questionnaire- will be used to assess participants' knowledge about their AAF condition. The scale consists of a total of 16 items and 3 sub-dimensions. The lowest score to be obtained from the scale is "0" and the highest score is "16". The higher the score obtained from the scale, the higher the patient's level of knowledge.
The University of Toronto Atrial Fibrillation Severity Scale | The measurement will be done at the beginning of the study (day 0) and at the end of the 12th week.
  The University of Toronto Atrial Fibrillation Severity Scale is a scale that will be used to assess the severity of AF-specific disease, the burden it creates in individuals and the frequency of AF episodes. The scale consists of 19 items and 3 sections. Higher scores indicate greater AF burden and more severe symptoms.
Effect of Atrial Fibrillation on Quality of Life Scale | The measurement will be done at the beginning of the study (day 0) and at the end of the 12th week.
  Effect of Atrial Fibrillation on Quality of Life Scale consists of four sub dimensions and 20 questions measuring the quality of life of patients with AF. Scoring of the scale ranges from 0 to 100 in general and sub-dimension scores. A score of zero indicates that quality of life is negatively affected.

SECONDARY OUTCOMES:
System Usability Scale-SUS | Measurement will be done at the end of the study (at the end of the 12th week).
  There are a total of 10 items in the System Usability Scale. Each item in the scale takes a value between 1 and 5. A total System Usability Scale score ranging from 0-100 is obtained. According to this score, systems or interfaces can be evaluated in terms of usability. The higher the score, the more usable the system is.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital Cardiology Polyclinic, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allan KS, Aves T, Henry S, Banfield L, Victor JC, Dorian P, Healey JS, Andrade JG, Carroll SL, McGillion MH. Health-Related Quality of Life in Patients With Atrial Fibrillation Treated With Catheter Ablation or Antiarrhythmic Drug Therapy: A Systematic Review and Meta-analysis. CJC Open. 2020 Apr 2;2(4):286-295. doi: 10.1016/j.cjco.2020.03.013. eCollection 2020 Jul. PMID 32695978
- [Background] Guo Y, Chen Y, Lane DA, Liu L, Wang Y, Lip GYH. Mobile Health Technology for Atrial Fibrillation Management Integrating Decision Support, Education, and Patient Involvement: mAF App Trial. Am J Med. 2017 Dec;130(12):1388-1396.e6. doi: 10.1016/j.amjmed.2017.07.003. Epub 2017 Aug 26. PMID 28847546
- [Background] Smigorowsky MJ, Norris CM, McMurtry MS, Tsuyuki RT. Measuring the effect of nurse practitioner (NP)-led care on health-related quality of life in adult patients with atrial fibrillation: study protocol for a randomized controlled trial. Trials. 2017 Aug 3;18(1):364. doi: 10.1186/s13063-017-2111-4. PMID 28774317
- [Background] Palm P, Qvist I, Rasmussen TB, Christensen SW, Hakonsen SJ, Risom SS. Educational interventions to improve outcomes in patients with atrial fibrillation-a systematic review. Int J Clin Pract. 2020 Nov;74(11):e13629. doi: 10.1111/ijcp.13629. Epub 2020 Sep 7. PMID 32726511
- [Background] Pearsons A, Hanson CL, Gallagher R, O'Carroll RE, Khonsari S, Hanley J, Strachan FE, Mills NL, Quinn TJ, McKinstry B, McHale S, Stewart S, Zhang M, O'Connor S, Neubeck L. Atrial fibrillation self-management: a mobile telephone app scoping review and content analysis. Eur J Cardiovasc Nurs. 2021 May 22;20(4):305-314. doi: 10.1093/eurjcn/zvaa014. PMID 33620473
- [Background] Willems S, Borof K, Brandes A, Breithardt G, Camm AJ, Crijns HJGM, Eckardt L, Gessler N, Goette A, Haegeli LM, Heidbuchel H, Kautzner J, Ng GA, Schnabel RB, Suling A, Szumowski L, Themistoclakis S, Vardas P, van Gelder IC, Wegscheider K, Kirchhof P. Systematic, early rhythm control strategy for atrial fibrillation in patients with or without symptoms: the EAST-AFNET 4 trial. Eur Heart J. 2022 Mar 21;43(12):1219-1230. doi: 10.1093/eurheartj/ehab593. PMID 34447995
- [Background] Joglar JA, Chung MK, Armbruster AL, Benjamin EJ, Chyou JY, Cronin EM, Deswal A, Eckhardt LL, Goldberger ZD, Gopinathannair R, Gorenek B, Hess PL, Hlatky M, Hogan G, Ibeh C, Indik JH, Kido K, Kusumoto F, Link MS, Linta KT, Marcus GM, McCarthy PM, Patel N, Patton KK, Perez MV, Piccini JP, Russo AM, Sanders P, Streur MM, Thomas KL, Times S, Tisdale JE, Valente AM, Van Wagoner DR; Peer Review Committee Members. 2023 ACC/AHA/ACCP/HRS Guideline for the Diagnosis and Management of Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jan 2;149(1):e1-e156. doi: 10.1161/CIR.0000000000001193. Epub 2023 Nov 30. PMID 38033089
- [Background] Boriani G, Vitolo M, Diemberger I, Proietti M, Valenti AC, Malavasi VL, Lip GYH. Optimizing indices of atrial fibrillation susceptibility and burden to evaluate atrial fibrillation severity, risk and outcomes. Cardiovasc Res. 2021 Jun 16;117(7):1-21. doi: 10.1093/cvr/cvab147. PMID 33913486
- [Background] Van Gelder IC, Rienstra M, Bunting KV, Casado-Arroyo R, Caso V, Crijns HJGM, De Potter TJR, Dwight J, Guasti L, Hanke T, Jaarsma T, Lettino M, Lochen ML, Lumbers RT, Maesen B, Molgaard I, Rosano GMC, Sanders P, Schnabel RB, Suwalski P, Svennberg E, Tamargo J, Tica O, Traykov V, Tzeis S, Kotecha D; ESC Scientific Document Group. 2024 ESC Guidelines for the management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2024 Sep 29;45(36):3314-3414. doi: 10.1093/eurheartj/ehae176. No abstract available. PMID 39210723
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://www.heart.org/en/health-topics/atrial-fibrillation
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://www.afibmatters.org/
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://www.cdc.gov/heart-disease/about/atrial-fibrillation.html
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://www.nhlbi.nih.gov/health/atrial-fibrillation
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://www.heartfoundation.org.au/your-heart/atrial-fibrillation
- See also: In the study, the educational content of the application developed for participants diagnosed with Atrial Fibrillation (M-AFEP, Mobile-Atrial Fibrillation Education Program) was used as a resource in the creation of the content. — https://tkd.org.tr/kardiyobil/